CLINICAL TRIAL: NCT05400044
Title: Assessment of Bone Quality and Quantity for Three Dimensional Bone Augmentation for Maxilla Using Patient Specific Titanium Meshes Loaded With Bone Marrow Aspirate Mixed With Xenograft Versus Xenograft Mixed With Autografts Only: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa, Mr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1222
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Atrophic Maxilla
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone marrow aspirate mixed with xenograft (Experimental)
  Interventions: Procedure: Three dimensional maxillary bone augmentation
- xenograft mixed with autografts only: (Active Comparator)
  Interventions: Procedure: Three dimensional maxillary bone augmentation

INTERVENTIONS:
Procedure: Three dimensional maxillary bone augmentation — mixing of bone marrow aspirate concentrate with xenograft to show the bone quality and bone gain compared to the xenografts mixed with autografts

SUMMARY:
Assessment of bone quality and quantity for three dimensional bone augmentation for maxilla using titanium meshes loaded with bone marrow aspirate mixed with xenograft versus xenograft mixed with autografts only

ELIGIBILITY:
Inclusion Criteria:

* Patients are free from any systemic conditions and bone metabolic diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.

  * Edentulous anterior or posterior maxilla with deficient alveolar ridge that is less than 5 mm measured from the crest of the alveolar ridge to the nasal or maxillary sinus and less than 4mm in buccolingual width.
  * The minimum number of missing teeth in the alveolar ridge is two adjacent teeth.

Exclusion Criteria:

* Intra-bony lesions (e.g. cysts) or infections (e.g. abscess) that may retard the osteotomy healing.

  * Previous grafting procedures in the edentulous area.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric bone analysis | 4 months
  ratio of mineralized tissue to non mineralized tissue

SECONDARY OUTCOMES:
Alveolar ridge vertical bone and horizontal bone gain | 4 months
  Gain measured in millimeters on a cone beam computed tomograpghy

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided